CLINICAL TRIAL: NCT04000100
Title: Effect OF Adding Neostigmine to Bupivacaine for Ultrasound Guided Supraclavicular Brachial Plexus Block in Forearm Surgeries
Brief Title: Neostigmine for Ultrasound Guided Supraclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ABEER HASSANIN (Other)
Responsible Party: Sponsor-Investigator, ABEER HASSANIN, Assistant Professor, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 72-7-2018
Record Dates: First submitted 2019-06-14; First posted 2019-06-27 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Postoperative Pain
Keywords: Neostigmine; Bupivacaine; Supraclavicular brachial plexus block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): This group received supraclavicular block using 25mL of 0. 5% bupivacaine and 1 mL normal saline
  Interventions: Procedure: ultrasound- guided supraclavicular brachial plexus block
- Neostigmine group (Active Comparator): This group received 25 mL 0. 5% bupivacaine and 1 mL neostigmine (0.5 mg)
  Interventions: Procedure: ultrasound- guided supraclavicular brachial plexus block

INTERVENTIONS:
Procedure: ultrasound- guided supraclavicular brachial plexus block — Patient lie down supine with head turned 45 degrees to the contralateral side and ipsilateral arm adducted gently by the assistant and the shoulder kept down with flexed elbow.
  After sterile preparation of the skin and the ultrasound probe (12 MHz probe) were used, the brachial plexus was visualized by placing the transducer in the sagittal plane in the supraclavicular fossa behind the middle-third of the clavicle. Two distinct appearances of the brachial plexus was seen at the supraclavicular region, it either appeared as 3 hypoechoic circles with hyperechoic outer rings or as a grape like cluster of 5 to 6 hypoechoic circles, located lateral and superior to the subclavian artery between the anterior and middle scalene muscles at the lower cervical region figure

SUMMARY:
Patients were randomly allocated into Two equal study groups each contain (40) patients : Patients in Group A received supraclavicular block using 25mL of 0. 5% bupivacaine and 1 mL normal saline and patients in Group B received 25 mL 0. 5% bupivacaine and 1 mL neostigmine (0.5 mg).

The investigators found that neostigmine when used as an adjuvant to bupivacaine in ultrasound guided supraclavicular brachial plexus block has advantage over bupivacaine alone especially in the quality of sensory block and provide safe and effective post-operative analgesia in patients undergoing forearm surgeries

DETAILED DESCRIPTION:
All patients were assessed with regards to:

Hemodynamics (heart rate, Bp) and oxygen saturation were recorded preoperatively just before the block as a baseline value, immediately after the block 5, 20, 30,40,45 , 60 minutes during the operative time and 1, 2, 4, 6, 9 and 12 hours after end of operation.

Onset time of sensory block, Onset time of motor block, Duration of sensory block, and Duration of motor block.

Pain assessment using a scoring system based on the visual analogue pain scale(VAS) measured at the following time intervals 0, 2, 4, 6, 9, 12 and 24 post operatively, time to first analgesic requirement (in hours) and total analgesic consumption was monitored in the two groups for 24 hours in ward.

The incidence of adverse effects whether related to the drugs used in the technique or related to the technique itself were recorded.

The results of this study found that demographic (age, sex, weight and ASA classification and surgical duration were statistically insignificant between the two groups.

Hemodynamics (HR and Bp) were statistically significant between the groups .They were lower in Neostigmine groups.

As regard onset of sensory and motor block were clinically and significantly earlier in group B than group A ( p < 0,05) and the same for duration of sensory and motor block were clinically and significantly longer in group B than in group A ( P < 0,05 ). Regarding Visual Analogue Pain Scale (VAS), while comparing the two groups, the differences were significant at 9 and 12 hours after surgery for the favor of the neostigmine groups . The time to first analgesic request was significantly longer in group B than group A.

ELIGIBILITY:
Inclusion Criteria:

1. ASA ( I-II)
2. Age: from ≥18 years
3. Sex: male or female
4. type of operation : Forearm Orthopedic surgeries
5. Type of anaesthesia : supraclavicular brachial plexus block
6. Duration of operation : 60-90 min

Exclusion Criteria:

1. Patient refusal for the procedure
2. Any bleeding tendency
3. Neurological deficits involving brachial plexus
4. Patients with allergy to local anesthetics
5. Local infection at the site of injection
6. Patients on any sedatives or antipsychotics
7. Body mass index >35.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
The onset of sensory blockade | Every 2 minutes for 30 minutes
  Onset time for sensory block was defined as the time interval between the end of local anesthetic administration untill complete sensory block by minutes
The onset of motor blockade | Every 2 minutes for 30 minutes
  Onset time for motor block was defined as the time interval between the end of local anesthetic administration until complete motor block by minutes
Duration of sensory blockade | Every 1 hour for 24 hours
  Duration of sensory block was defined as the time interval between the complete sensory block and complete resolution of anesthesia on all the nerves by hours
Duration of motor blockade | Every 1 hour for 24 hours
  the time interval from complete motor block to complete recovery of motor function of hand and forearm by hours

SECONDARY OUTCOMES:
Duration of analgesia (first request for analgesic) | Every 30 minutes for 4 hours then every 2 hours for 24 hours
  The time from local anesthetic administration to the patient's first request for analgesic medication by hours
Visual analogue pain score | 2,4,6,8,12,16,20 and 24 hours postoperative
  Pain intensity was assessed using Visual analogue pain score. The Visual analogue pain score is consisted of a straight ,vertical 10-cm line; the bottom point represented "no pain"=(0 cm) and the top "the worst pain you could ever have =(10 cm)

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim Abbas, MD, Study Director — faculty of medicine
Locations (1):
- Minya university hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data can be shared
Supporting Information: Study Protocol, SAP
Time Frame: From now
Access Criteria: abeerhassanin@yahoo.com